CLINICAL TRIAL: NCT05457504
Title: Blood Pressure Monitoring in Postpartum Women at Risk of Hypertension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Ilona T. Goldfarb, M.D., Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2021P003705
Record Dates: First submitted 2022-07-11; First posted 2022-07-14 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Hypertension in Pregnancy; Preeclampsia; Gestational Hypertension; Chronic Hypertension With Pre-Eclampsia; Hypertension Complicating Pregnancy, Childbirth, and the Puerperium
MeSH Terms: conditions — Hypertension, Pregnancy-Induced; Pre-Eclampsia

STUDY DESIGN:
Intervention Model Description: In this study, we are testing different strategies to help women decrease issues with hypertension in the postpartum period. Participants may or may not undergo some of the following study procedures:
  * Frequent blood pressure monitoring and feedback
  * Receive information related to blood pressure measurement, heart disease prevention, etc.
  * Regular blood pressure monitoring and advice regarding changes in medications.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental)
  Interventions: Behavioral: Remote blood pressure monitoring
- Usual Care (Placebo Comparator)
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Remote blood pressure monitoring — Participants assigned to this arm will participate in the experimental intervention
  Arms: Experimental
Behavioral: Usual Care — Participants assigned to this arm will participate in a placebo intervention
  Arms: Usual Care

SUMMARY:
Cardiovascular disease and hypertensive disorders of pregnancy (HDP) are the leading causes of maternal morbidity and mortality in the United States. Postpartum, in office care has demonstrated to be an insufficient model of hypertensive management postpartum, largely due to barriers that women face in accessing in office care, with stark racial disparities in access. The care of postpartum patients with HDP following delivery is made up of either a single postpartum visit at 6 weeks postpartum or a fragmented and non-standardized series of in-person appointments depending on the patients' medical complications and the clinicians' experience. Further, current society guidelines outline inpatient thresholds for initiation of antihypertensive medication but do not provide recommendations for titration thereafter. The proposed study will investigate the acceptability and effectiveness of an algorithm-based, outpatient treatment model for the management of postpartum hypertension utilizing an asynchronous text-based platform as compared to the standard of care for postpartum women with a diagnosis of Hypertensive disorder of pregnancy at Massachusetts General Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Diagnosis of gestational hypertension (Systolic Blood Pressure (SBP)≥140 or Diastolic Blood Pressure (DBP) ≥90 on at least two occasions at least 4 hours apart after 20 weeks gestation in previously normotensive women) and or preeclampsia (SBP≥140 or DBP ≥90, proteinuria with or without symptoms of preeclampsia (headache, vision changes, right upper quadrant pain), and presentation of symptoms/lab abnormalities but no proteinuria)
* English and Spanish-speaking
* Delivering at Massachusetts General Hospital

Exclusion Criteria:

* Chronic hypertension or underlying cardiovascular disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Percent of patients who are normotensive at 6 weeks postpartum by American College of Cardiology (ACC)/American Heart Association (AHA) guidelines | 6 weeks
  Percent of patients who are normotensive at 6 weeks postpartum by ACC/AHA guidelines (>130/80) in each treatment group

SECONDARY OUTCOMES:
Percent of patients who are normotensive at 6 weeks postpartum by American College of Obstetricians and Gynecologists (ACOG) guidelines | 6 weeks
  Percent of patients who are normotensive at 6 weeks postpartum by ACOG guidelines (>140/90) in each treatment group
Frequency of Hospital readmission | 6 weeks
  Frequency of Hospital readmission in the first 6 weeks postpartum in each treatment group
Number of medication titrations | 6 weeks
  Mean number of medication titrations by patient in the first 6 postpartum weeks in each treatment group
Adherence with scheduled outpatient clinical appointments | 6 months
  Percent of scheduled outpatient clinical appointments attended by patients in the first 6 postpartum months in each treatment group
Establishment of care with a primary care doctor | 1 year
  Percent of patients who attend a primary care doctor visit in the first postpartum year in each treatment group